CLINICAL TRIAL: NCT06662747
Title: Vaginal Microbiome Research Consortium for Africa - Pilot
Brief Title: Vaginal Microbiome Research Consortium for Africa
Acronym: VMRC4Africa
Status: Recruiting | Type: Observational
Sponsor: University of Cape Town (Other)
Collaborators: Desmond Tutu HIV Foundation (Other); Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Jo-An Passmore, Professor, University of Cape Town
Other Study IDs: INV-037612
Record Dates: First submitted 2024-07-24; First posted 2024-10-29 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Swab 1 - 1x Valvo vaginal swab for STI testing (this may be self-collected) Swab 2 - 1x High-vaginal wall for storage Swab 3 - 1x lateral vaginal wall swab to be applied to pH indicator and rolled on a glass slide for Nugent scoring Swab 4 - 1x lateral vaginal wall swab for qPCR and 16S rRNA (bacterial) & ITS (fungal) amplicon sequencing (Molecular transport medium [Qiagen]) Swab 5 - 1x Lateral wall swab for culture (Amies-based transport solution, eg E-Swab [Copan]) (culture)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy: Cervicovaginal microbiota, mycobiota, and HPV prevalence, and identify women with stable Lactobacillus-dominated microbiota, with no STIs and no evidence of genital inflammation.
  Interventions: Diagnostic Test: None - observational study only

INTERVENTIONS:
Diagnostic Test: None - observational study only — No interventions, diagnostics tests for HIV, pregnancy, STIs and BV only

SUMMARY:
1. To characterise vaginal microbial community dynamics (bacterial and fungal) from different geographies in Africa to understand the microbial diversity that occurs in women with stable L. crispatus-dominant versus unstable vaginal microbiota.
2. To identify vaginal communities associated with low levels of inflammation in women from different geographies in Africa
3. To examine prevalence and diversity of HPV types circulating in the different geographies and their interaction with the vaginal microbiota
4. To create a biobank of stored samples that can be used in future studies and for the isolation of regionally representative bacterial strains.

DETAILED DESCRIPTION:
This investment forms part of the BMGF Calestous Juma Scientific Leadership (CJSL) Fellowship to Dr Jo-Ann Passmore, to pilot VMRC4Africa and establish a collaborative regional network with African partners and Centres of Excellence with capacity and expertise to conduct clinical trials and vaginal microbiome research in Africa. With this CJSL Fellowship investment, Dr Passmore and her collaborators aim to enrol parallel cohorts of women from two sites in two African countries (South Africa: Desmond Tutu HIV Foundation [DTHF] and Kenya Medical Research Institute [KEMRI]) to evaluate detailed temporal fluctuations in vaginal microbiota in young, generally healthy women from Southern and Eastern Africa. These parallel cohorts will be intensively followed for 10 weeks, to create detailed profiles of vaginal microbial community state types (CSTs; by 16S rRNA gene sequencing) and fungal communities [by internal transcribed spacer (ITS) sequencing], to identify women with stable Lactobacillus-dominated microbiota, with no evidence of genital inflammation. Through the establishment of an "African vaginal microbiome biorepository", the intention will be to create a biobank from which to ultimately select geographically diverse Lactobacillus crispatus strains with health promoting characteristics that can be co-formulated into live biotherapeutic products (LBPs) to treat bacterial vaginosis (BV) for women globally.

ELIGIBILITY:
Inclusion Criteria:

* Female at birth
* Willing and able to provide informed consent for screening and cognitive ability to understand sampling procedures
* Not pregnant
* HIV negative on testing performed by study staff
* 18-40 years old
* Planning to stay in the area for the next 10 weeks
* Able and willing to provide adequate locator information for study retention purposes
* Willing and able to return for all 3 nurse visits and return self-swabs to the clinic weekly
* Sexually active for the last 3 months defined as penetrative penile-vaginal intercourse at least once in the last 3 months

Exclusion Criteria:

* Male at birth
* Not willing to provide consent
* Pregnant or actively trying to conceive/become pregnant in the next 10 weeks
* Living with HIV or untreated STIs (CT, NG, TV) or bacterial vaginosis (Nugent > 3)
* Currently taking antibiotics or having been on antibiotic treatment in the previous four weeks
* <18 or >40 years old
* On chronic disease management for gynaecological conditions
* Any medical condition or other factors which would preclude study participation as per principal Investigator's or designee's decision, including but not limited to cancer of the cervix
* Any mental health condition which, in the opinion of the investigator, would preclude comprehension of informed consent, or preclude study participation
* Currently enrolled on any other study prohibiting co-enrolment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female at birth
Study Population: Participants will be recruited via the CRS standard recruiting process. Participants will be informed about the study via social media, flyers and posters. Each site will use a variety of recruitment approaches that works best for the local setting.
  Recruitment may be conducted through the following possible approaches: community events and mobilisation, partnerships with appropriate programs and via popular social media platforms. Recruitment materials will educate women about HIV, sexual health, and risks in their community, the effectiveness of PrEP for HIV prevention, and the benefits of HIV prevention services. Recruitment will occur over approximately 12 months.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Geographic Insights into Vaginal Microbial Diversity: Characterizing Bacterial and Fungal Community Dynamics in African Women with Stable L. crispatus-Dominated vs. Unstable Microbiota. | 5 years
  The study measures the dynamics of vaginal microbial communities (bacterial and fungal) across different African geographies in women with stable L. crispatus-dominant and unstable microbiota. Specific measurements include the recovery of bacterial and fungal DNA through DNA extraction methods. For bacterial profiling, the analysis includes the use of 16S rRNA gene sequencing targeting the V3-V4 variable regions, while fungal diversity, specifically Candida species, is assessed via Internal Transcribed Spacer (ITS) sequencing. The sequencing data is processed using bioinformatics tools such as QIIME2 and DADA2 for quality control, filtering, and taxonomic assignment. Alpha (within-sample) and beta (between-sample) diversity are measured using metrics including the Shannon index and Bray-Curtis dissimilarity. Additionally, multivariate techniques such as NMDS and PCA are employed to visualize community structures and differences.
Explore Vaginal Microbiome Profiles and Their Association with Low Inflammatory States in Women Across Diverse African Geographies. | 3 years
  This study measures vaginal microbial communities associated with low inflammation levels in women across various African geographies. The assessment includes the prevalence of HPV types in different regions, evaluated through statistical tests such as Chi-square and logistic regression to determine geographic variations. The composition of the vaginal microbiota will be analyzed using bioinformatics techniques to report alpha (within-sample) and beta (between-sample) diversity metrics. Significant variations in microbiota profiles across regions will be identified using ANOSIM and PERMANOVA statistical methods. Correlations between specific HPV types and microbiota profiles will be quantified using Spearman or Pearson correlation coefficients to assess their interactions.
Geographic Variation in HPV Type Prevalence and Divers. | 5 years
  This study will measure HPV type prevalence and diversity across various geographies, as well as its interaction with vaginal microbiota. HPV prevalence will be quantified using molecular methods including PCR and next-generation sequencing (NGS) for DNA detection and type analysis. Vaginal microbiota will be profiled by extracting microbial DNA from swabs, followed by 16S rRNA gene sequencing or metagenomics.
  The outcome measures include the calculation of HPV prevalence and diversity, utilizing metrics such as the Shannon index. Additional outcome measures involve statistical analysis to characterize relationships between HPV types and microbiota composition, as well as correlation analysis to identify links between specific HPV types and microbial species. This analysis aims to clarify the role of the microbial community in HPV infection and persistence, with a focus on identifying potential protective effects of specific microbiota profiles.
Establishment of a Regional Biobank | 4 years
  Create a biobank of stored samples that can be used in future studies and for the isolation of regionally representative bacterial strains.

CONTACTS AND LOCATIONS:
Overall Officials: Brian R Kullin, PhD, Study Director — Research Officer
Locations (2):
- KEMRI, Kisumu, Kisumu County, Kenya
- Desmond Tutu Health Foundation, Cape Town, Western Cape, South Africa